CLINICAL TRIAL: NCT06901986
Title: Health Benefits of Montmorency Tart Cherry Juice Supplementation in Adults with Mild to Moderate Crohn's Disease.
Brief Title: Health Benefits of Tart Cherry in Crohn's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire (Other)
Collaborators: University of Hertfordshire (Other)
Responsible Party: Principal Investigator, Jonathan Sinclair, Professor, University of Central Lancashire
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tart cherry Crohn's disease
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Crohn Disease (CD)
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Montmorency tart cherry juice (Experimental): Dietary Supplement: Montmorency tart cherry Description: US grown Montmorency tart cherry 60ml per day for 6 weeks.
  Interventions: Dietary Supplement: Montmorency tart cherry
- Placebo (Placebo Comparator): Taste matched placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Montmorency tart cherry — Montmorency tart cherry 60ml per day for 6 weeks.
  Arms: Montmorency tart cherry juice
Dietary Supplement: Placebo — Taste matched placebo.
  Arms: Placebo

SUMMARY:
Crohn's disease (CD) is a long-term inflammatory condition of the digestive tract. People with CD often experience unpredictable and debilitating symptoms, including abdominal pain, diarrhea, and fatigue. Additionally, they require long-term treatment, which is often associated with frequent negative effects, the need for surgery, and hospitalizations. As a result, individuals with CD report a lower health-related quality of life (HRQOL) compared to healthy individuals.

The most common medication for inflammatory bowel disease is a strong immunosuppressant, which was identified in 2017 as the most expensive medication prescribed in NHS hospitals. Unfortunately, biologics have significant side effects, and reducing the reliance on them could benefit both the NHS by lowering costs and patients by minimizing unwanted side effects.

Supplementation with Montmorency tart cherry juice may offer a simple, safe, and cost-effective intervention for improving symptoms in individuals with CD. This is due to its potential to naturally reduce inflammation in the digestive system, thereby alleviating symptoms. Research in animal models has shown potential improvements in physiological responses with similar supplements, including blueberries, black raspberries, and Montmorency tart cherries, though only one study in human participants has explored bilberry supplementation.

Despite Montmorency tart cherries having superior anthocyanin concentrations compared to other berries, dietary interventions using tart cherry supplementation for CD have not been explored in human participants. The primary aim of the proposed investigation is to conduct a placebo-controlled randomized trial to examine whether Montmorency tart cherry juice supplementation can provide symptom relief and improve health-related well-being in individuals with mild to moderately active CD, as well as to understand the biological mechanisms underlying any observed symptom changes.

ELIGIBILITY:
Inclusion Criteria:

* An established diagnosis of CDfor at least 6 months
* Current mild to moderate disease activity
* Age between 18 and 65 years
* Stable use of medication for at least 3 months respectively.

Exclusion Criteria:

* Diabetes
* HIV
* Hepatitis B and C infection
* Abscesses
* Unstable medical conditions that would likely prevent the subject from completing the study
* Food allergies to cherries.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Bowel Disease Quality of Life Questionnaire | This parameter will be examined at baseline.
  The scale has 32 items scored on a 7-point Likert scale, ranging from 1 (worst health) to 7 (best health).
Inflammatory Bowel Disease Quality of Life Questionnaire | This parameter will be examined at 6 weeks
  The scale has 32 items scored on a 7-point Likert scale, ranging from 1 (worst health) to 7 (best health).

SECONDARY OUTCOMES:
Simple clinical colitis activity index | This parameter will be examined at baseline.
  The calculated score ranges from 0 to 19, where active disease is a score of 5 or higher.
Hospital anxiety and depression scale | This parameter will be examined at 6 weeks
  The Hospital Anxiety and Depression Scale measures anxiety and depression in patients. A higher score indicates greater anxiety and depression.
European Quality of Life Scale | This parameter will be examined at baseline.
  The European Quality of Life Scale is an instrument for measuring quality of life across patient groups and cultures and is conceptually distinct from health status or other causal indicators of quality of life. A higher score indicates higher quality of life.
European Quality of Life Scale | This parameter will be examined at 6 weeks
  The European Quality of Life Scale is an instrument for measuring quality of life across patient groups and cultures and is conceptually distinct from health status or other causal indicators of quality of life. A higher score indicates higher quality of life.
International Physical Activity Questionnaire - Short Form | This parameter will be examined at baseline.
  The International Physical Activity Questionnaire - Short Form (IPAQ-SF) addresses the number of days and time spent on physical activity in moderate intensity, vigorous intensity and walking of at least 10-min duration the last 7 days, and also includes time spent sitting on weekdays the last 7 days. The IPAQ-SF sum score is expressed in physical activity Metabolic Equivalent of Task minutes per day or week.
International Physical Activity Questionnaire - Short Form | This parameter will be examined at 6 weeks
  The International Physical Activity Questionnaire - Short Form (IPAQ-SF) addresses the number of days and time spent on physical activity in moderate intensity, vigorous intensity and walking of at least 10-min duration the last 7 days, and also includes time spent sitting on weekdays the last 7 days. The IPAQ-SF sum score is expressed in physical activity Metabolic Equivalent of Task minutes per day or week.
IBD Fatigue Scale | This parameter will be examined at baseline
  The IBD Fatigue Scale is comprised of two components. Part 1 the questionnaire will identify fatigue, its severity, frequency and duration and scores range from 0-20 with a higher score meaning greater fatigue. Part 2 assesses the perceived impact of fatigue on your daily activities and scores range from 0-120 with a higher score meaning greater perceived impact.
IBD Fatigue Scale | This parameter will be examined at 6 weeks
  The IBD Fatigue Scale is comprised of two components. Part 1 the questionnaire will identify fatigue, its severity, frequency and duration and scores range from 0-20 with a higher score meaning greater fatigue. Part 2 assesses the perceived impact of fatigue on your daily activities and scores range from 0-120 with a higher score meaning greater perceived impact.
Faecal calprotectin | This parameter will be examined at baseline
  Faecal calprotectin is a stool test that measures the protein calprotectin, released by neutrophils during inflammation, to assess gut inflammation.
Faecal calprotectin | This parameter will be examined at 6 weeks
  Faecal calprotectin is a stool test that measures the protein calprotectin, released by neutrophils during inflammation, to assess gut inflammation.
Gut microbiome | This parameter will be examined at baseline
  The gut microbiome in individuals with IBD differs significantly from that of healthy individuals, with a reduction in beneficial bacteria and an increase in potentially harmful bacteria.
Faecal calprotectin | This parameter will be examined at 6 weeks
  The gut microbiome in individuals with IBD differs significantly from that of healthy individuals, with a reduction in beneficial bacteria and an increase in potentially harmful bacteria.

IPD SHARING:
Plan to Share IPD: No